CLINICAL TRIAL: NCT03728166
Title: Randomized Controlled Trial of Computerized Decision Support for Prevention of Venous Thromboembolism in Hospitalized Medical Patients Across the Continuum of Care (DC-eALERT)
Brief Title: Computerized Decision Support for Prevention of VTE in Hospitalized Medical Patients Across the Continuum of Care (DC-eALERT)
Acronym: DC-eALERT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Portola Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Gregory Piazza, MD, MS, Associate Director, Thrombosis Research Group, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2018P001727
Record Dates: First submitted 2018-10-30; First posted 2018-11-01 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Venous Thromboembolism
Keywords: venous thromboembolism; prevention; medical patients; hospital discharge
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Intervention Model Description: U.S.-based, single-center, randomized controlled trial
Who Masked: Participant
Masking Description: Investigators will randomize patients by Attending Physician ID# to minimize the influence of an alert effect on the care of patients not randomized to the alert group but who have the same Attending Physician (thereby reducing what is called the "cluster-effect"). While investigators will randomize patients by Attending Physician of Record to minimize cluster-effect, the observational unit will be the patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Alert (Experimental): On-screen electronic alert that notifies the provider about the increased risk for VTE after discharge and indication for thromboprophylaxis will be issued 48 hours after admission. This first on-screen electronic alert will provide the clinician with the opportunity to consider extended-duration, post-discharge thromboprophylaxis and start any required processes for prior authorization or medication coverage. The provider then will be given on-screen options to either order thromboprophylaxis (betrixaban or low-molecular weight heparin for 35 days) from a "Extended-Duration VTE Prevention" order template, follow a link to evidence-based practice guidelines, or defer prescribing extended-duration, post-discharge thromboprophylaxis.
  Interventions: Behavioral: Electronic alert
- No Alert (No Intervention): No notification to the provider.

INTERVENTIONS:
Behavioral: Electronic alert — On-screen electronic alert that notifies the provider about the increased risk for VTE after discharge and indication for thromboprophylaxis will be issued 48 hours after admission. This first on-screen electronic alert will provide the clinician with the opportunity to consider extended-duration, post-discharge thromboprophylaxis and start any required processes for prior authorization or medication coverage. The provider then will be given on-screen options to either order thromboprophylaxis (betrixaban or low-molecular weight heparin for 35 days) from a "Extended-Duration VTE Prevention" order template, follow a link to evidence-based practice guidelines, or defer prescribing extended-duration, post-discharge thromboprophylaxis.
  Arms: Alert

SUMMARY:
Hospitalized medical patients have an increased risk of venous thromboembolism (VTE) across the continuum of care, including after hospital discharge. In the APEX Trial of hospitalized patients with acute medical illness, extended-duration post-discharge thromboprophylaxis with oral betrixaban reduced the frequency of asymptomatic proximal deep venous thrombosis (DVT), symptomatic proximal or distal DVT, symptomatic nonfatal pulmonary embolism (PE), or VTE-related death compared with short-duration enoxaparin. Obstacles to integration of these data in the hospitalized Medical Service patient population, including failure to identify at-risk patients, educational gaps in strategies for VTE prevention after discharge, and medication nonadherence, can be overcome with alert-based computerized decision support. This study is a single-center, 400-patient, randomized controlled trial of an EPIC Best Practice Advisory (BPA; alert-based computerized decision support tool) to increase prescription of extended-duration post-discharge thromboprophylaxis and decrease symptomatic VTE in high-risk patients hospitalized with medical illness.

Specific Aim #1: To determine the impact of electronic alert-based CDS (EPIC Best Practice Advisory [BPA]) on prescription of extended-duration post-discharge thromboprophylaxis in high-risk patients hospitalized with medical illness who are not being prescribed any prophylactic anticoagulation for VTE prevention after discharge.

Specific Aim #2: To estimate the impact of electronic alert-based CDS (EPIC BPA) on the frequency of symptomatic VTE in high-risk patients hospitalized with medical illness who are not being prescribed any prophylactic anticoagulation for VTE prevention after discharge.

DETAILED DESCRIPTION:
Design: U.S.-based, single-center, randomized controlled trial

Background: Hospitalized medical patients have an increased risk of venous thromboembolism (VTE) across the continuum of care (from before admission to after discharge). In the APEX Trial of 7513 hospitalized patients with acute medical illness, reduced mobility, and risk factors for VTE, extended-duration post-discharge thromboprophylaxis with oral betrixaban for 35 to 42 days reduced the frequency of asymptomatic proximal deep venous thrombosis (DVT), symptomatic proximal or distal DVT, symptomatic nonfatal pulmonary embolism (PE), or VTE-related death by 24% in the overall study population compared with 10-14 days of enoxaparin. The integration of oral betrixaban with a computerized decision support (CDS) tool has the potential to increase the appropriate prescription of extended-duration post-discharge thromboprophylaxis in high-risk patients hospitalized with medical illness.

Study Design: 400-patient U.S.-based single-center Quality Improvement Initiative in the form of a randomized controlled trial focused on the feasibility of implementation of this electronic alert-based CDS (EPIC BPA) (Figure 1). The allocation ratio will be 1:1 for an electronic alert-based CDS (EPIC BPA) notification versus no notification.

Study Population: Patients are eligible if they are ≥40 years of age, are hospitalized for acute medical illness (heart failure, respiratory failure, infectious disease, rheumatic disease, or ischemic stroke), have reduced mobility, and have one additional risk factor for VTE:

1. Age ≥60
2. Prior VTE
3. History of cancer

Eligible patients are not prescribed thromboprophylaxis at hospital discharge.

Intervention: An EPIC Electronic Health Record (EHR) Best Practice Advisory (BPA) will identify patients hospitalized with medical illness who are not ordered for extended-duration, post-discharge thromboprophylaxis 48 hours after admission. A first on-screen electronic alert will provide the clinician with the opportunity to consider extended-duration, post-discharge thromboprophylaxis and start any required processes for prior authorization or medication coverage. A second on-screen electronic alert will be issued if extended-duration, post-discharge thromboprophylaxis has still not been ordered that again notifies the provider about the increased risk for VTE after discharge and indication for thromboprophylaxis.

Primary Efficacy Outcome: Prescription of extended-duration post-discharge thromboprophylaxis. Investigators will review the order entry section of the Electronic Health Record (EPIC) to make this determination.

Secondary Efficacy Outcome: Frequency of symptomatic VTE at 90 days from randomization. Investigators will review the notes and diagnostic testing sections of the Electronic Health Record (EPIC) to make this determination. The proposed study will not be powered to show a difference in clinical events, such as symptomatic VTE, with the electronic alert-based CDS but will provide estimates from which to plan a possible subsequent multi-center trial.

Primary Safety Outcome: Major bleeding (as defined by the ISTH bleeding classification system) at 90 days from randomization. Investigators will review the notes and diagnostic testing sections of the Electronic Health Record (EPIC) to make this determination. The proposed study will not be powered to show a difference in clinical events, such as bleeding, with the electronic alert-based CDS but will provide estimates from which to plan a possible subsequent multi-center trial.

Follow-Up: Follow-up will consist of Electronic Health Record review at 90 days from randomization.

ELIGIBILITY:
Inclusion Criteria:

-≥40 years of age, are hospitalized for acute medical illness (heart failure, respiratory failure, infectious disease, rheumatic disease, or ischemic stroke), have reduced mobility, are not prescribed thromboprophylaxis at hospital discharge, and have one additional risk factor for VTE:

* Age ≥60
* Prior VTE OR
* History of cancer

Exclusion Criteria:

- Prescribed thromboprophylaxis at hospital discharge

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of prescription of extended-duration post-discharge thromboprophylaxis. | 90 days
  Investigators will review the order entry section of the Electronic Health Record (EPIC) to make this determination.

SECONDARY OUTCOMES:
Frequency of symptomatic VTE at 90 days from randomization. | 90 days
  Investigators will review the notes and diagnostic testing sections of the Electronic Health Record (EPIC) to make this determination. The proposed study will not be powered to show a difference in clinical events, such as symptomatic VTE, with the electronic alert-based CDS but will provide estimates from which to plan a possible subsequent multi-center trial.
Frequency of major bleeding (as defined by the ISTH bleeding classification system) at 90 days from randomization. | 90 days
  Investigators will review the notes and diagnostic testing sections of the Electronic Health Record (EPIC) to make this determination. The proposed study will not be powered to show a difference in clinical events, such as bleeding, with the electronic alert-based CDS but will provide estimates from which to plan a possible subsequent multi-center trial.
Frequency of all-cause mortality at 90 days | 90 days
  Any death confirmed by medical record
Frequency of all-cause rehospitalization at 90 days | 90 days
  Any rehospitalization confirmed by medical record

OTHER OUTCOMES:
Medication adherence | 35 days
  The proportion of patients who completed the 35-day course of post-discharge thromboprophylaxis.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Piazza, MD, MS, Principal Investigator — BWH
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cohen AT, Harrington RA, Goldhaber SZ, Hull RD, Wiens BL, Gold A, Hernandez AF, Gibson CM; APEX Investigators. Extended Thromboprophylaxis with Betrixaban in Acutely Ill Medical Patients. N Engl J Med. 2016 Aug 11;375(6):534-44. doi: 10.1056/NEJMoa1601747. Epub 2016 May 27. PMID 27232649